CLINICAL TRIAL: NCT03524001
Title: Bifocal Right Ventricular PAcing in Right Bundle Branch blocK and Heart Failure With Reduced Ejection Fraction
Brief Title: Bifocal Right Ventricular PAcing in Right Bundle Branch blocK and Heart Failure With Reduced Ejection Fraction. The Study Tests the Superiority of Right Ventricular Bifocal Stimulation Over VVI Implantable Defibrillator in Right Bundle Branch Block and Heart Failure.
Acronym: BiPARK-HF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Non superiority of treatment arm (and hypothesized inferiority) before completion of enrolling, at ad interim analysis
Sponsor: Azienda Ospedaliero Universitaria Maggiore della Carita (Other)
Responsible Party: Principal Investigator, Gabriele Dell'Era, Medical Doctor, Azienda Ospedaliero Universitaria Maggiore della Carita
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CE 194/17
Record Dates: First submitted 2018-04-18; First posted 2018-05-14 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Right Bundle-Branch Block; Heart Failure With Reduced Ejection Fraction; Bifocal Stimulation
MeSH Terms: conditions — Bundle-Branch Block

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bifocal stimulation (Active Comparator): Active comparator is represented by programming bifocal stimulation (bifocal DDD mode). Every patients will undergo crossover randomization (from bifocal DDD mode to VVI and vice versa).
  Interventions: Device: Compare VVi mode versus DDD bifocal stimulation through crossover randomization
- VVI 40 (Placebo Comparator): Placebo comparator is represented by programming the device in VVI mode 40/mins. Every patients will undergo crossover randomization (from VVI to bifocal DDD mode and vice versa).
  Interventions: Device: Compare VVi mode versus DDD bifocal stimulation through crossover randomization

INTERVENTIONS:
Device: Compare VVi mode versus DDD bifocal stimulation through crossover randomization — All patients undergo bifocal right ventricular resynchronization therapy: right atrial lead is implanted, whereas first ventricular lead is placed in His bundle area, and the second ventricular lead in the right ventricle apex.Then the leads are connected to CRT-D generator.After the implant, all devices are programmed in VVI mode. After the first 40±10 days (first f-up) patients are 1:1 randomized to VVI mode 40 beats/minute (placebo arm) or bifocal DDD-mode 60 beats/minute.After six months (second follow-up) a clinical and instrumental assessment equal to baseline is performed. Then arms cross-over is performed (from VVI-mode to bifocal DDD-mode and vice versa). At 12 months (end of follow-up) an evaluation equal to that performed at 6 months is assessed. Echocardiographic data are unravelled to the investigator that plans stimulation mode able to determine the best clinical improved.

SUMMARY:
RATIONALE:

Cardiac resynchronization therapy (CRT) is known to improve cardiac performance and to reduce morbidity and mortality in reduced-ejection fraction heart failure (HFrEF) despite optimal medical therapy (OMT). Several studies have shown that patients with with left bundle branch block (LBBB) respond favourably to CRT, whereas there is less certainty about non-LBBB morphology.

Specifically, whether patients with right bundle branch block (RBBB) and HFrEF benefit from CRT is unclear. Some studies suggest lack of favourable outcomes. It follows from this that VVI implantable defibrillator are implanted in most RBBB patients.On the other hand right ventricular bifocal stimulation could be useful as an alternative approach in patient with RBBB. It consists of two endocardial leads implanted in right ventricle. The first lead is implanted in His bundle area, and the second lead is in the right ventricle apex. In this way bifocal pacing could decrease the inter- and intraventricular delays, thus improving left ventricular hemodynamics. However no specifically randomized studies are designed to date.

PURPOSE:

To demonstrate the superiority of right ventricular bifocal stimulation over placebo (VVI implantable defibrillator) in RBBB and HFrEF despite OMT.

DESIGN Multicenter prospective randomized, double blind cross-over study. MASKING Investigator responsible for device programming is masked from having knowledge about clinical, functional, and echocardiographic data. On the other hand echocardiographist is masked from having knowledge about stimulation mode. Patients are masked from having knowledge about their clinical, functional, and device data.

POPULATION At least fifty patients would be enrolled. The enrollment period should be one year. Study overall duration should be two years.

ELIGIBILITY CRITERIA RBBB and HFrEF (left ventricular ejection fraction ≤35%) in sinus rhythm, in NYHA class II-III or ambulatory IV despite OMT.

EXCLUSION CRITERIA

-Refusal or withdrawal of informed consent.Renal failure (glomerular filtration rate ≤ 60 ml/min).Life expectancy < 12 months.Active neoplasm.Permanent atrial fibrillation.40 days following acute coronary syndrome.Atrio-ventricular block (from second degree AV block).Valvular heart disease with surgery indications.

PROTOCOL Each patient undergoes baseline assessment. Pharmacological therapy, hospitalization,NYHA functional class, QRS complex informations, type of heart disease and comorbidities are collected. Quality of life (QOL) is defined by Minnesota Living with Heart Failure questionnaire. Functional capacity is assessed by 6MWT (optionally by cardiopulmonary exercise test). Trans-thoracic echocardiogram is performed, analyzing: left-ventricle diameters and volumes, left-ventricle ejection fraction (LVEF), left atrial diameter and area, TAPSE,valvulopathy,systolic pulmonary artery pressure. All patients undergo bifocal right ventricular resynchronization therapy: right atrial lead is implanted, whereas the first ventricular lead is placed in His bundle area, and the second ventricular lead in the right ventricle apex. Then the leads are connected to the respective channels of a CRT-D generator.After the implant, all devices are programmed in VVI mode. After the first 40±10 days (first f-up) patients are 1:1 randomized to VVI mode 40 beats/minute (placebo arm) or bifocal DDD-mode 60 beats/minute (with VV delay 0 msec and optimal AV delay). After six months (second f-up) a clinical and instrumental assessment equal to baseline is performed, as well as devices electrical parameters control. Then arms cross-over is performed (from VVI-mode to bifocal DDD-mode and vice versa). At 12 months (end of follow-up) an evaluation equal to that performed at 6 months is assessed. Echocardiographic data are unravelled to the investigator responsible for device programming. In this way the stimulation mode able to determine the best clinical improved (VVI or bifocal DDD mode) is programmed and the study closes.

PRIMARY ENDPOINT The main assumption is that bifocal stimulation can increase of at least 20% the distance walked during 6MWT in respect of baseline and VVI-mode.The primary endpoint is the distance walked (expressed by meters) during 6MWT, as assessed at baseline, 6-months follow-up and 12 months follow up. Specifically changes in 6MWT observed during bifocal DDD-mode compared to baseline and to VVI mode would be significative if there is an increase of at least 20%.

SECONDARY ENDPOINT

Secondary endpoint is bifocal stimulation therapy response, defined by at least one of the following criteria, evaluated at baseline, 6-months follow-up and 12 months-follow-up in comparison to baseline and VVI mode:

NYHA functional class improvement; changes in 6MWT, defined by an increase in distance walked major or equal to 30%; LVEF improvement major or equal to 25%;Left ventricular telesystolic volume reduction major or equal to 15%

ELIGIBILITY:
Inclusion Criteria:

* Patients with RBBB and HFrEF (defined by left ventricular ejection fraction ≤35%) in sinus rhythm, who remain in NYHA class II-III or ambulatory NYHA class IV despite OMT.

Exclusion Criteria:

* Refusal or withdrawal of informed consent.
* Renal failure (defined by an estimated glomerular filtration rate ≤ 60 ml/min)
* Life expectancy < 12 months
* Active neoplasm
* Permanent atrial fibrillation
* 40 days following acute coronary syndrome
* Atrio-ventricular block (from second degree AV block)
* Valvular heart disease with surgery indications

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2022-06-27 (Actual); Study Completion 2022-07-10 (Actual)

PRIMARY OUTCOMES:
Change (expressed as a percentage) in distance walked during six-minute walk test (6MWT). 6MWT distance is expressed in meters | baseline, 6 months follow-up, 12 months follow-up
  the primary endpoint is the distance walked during 6MWT, expressed in meters. Specifically changes (expressed as a percentage) in 6MWT distance observed during bifocal DDD-mode compared to baseline and to VVI mode are registered and would be significative if there is an increase of at least 20%.

SECONDARY OUTCOMES:
New York Heart Association (NYHA) functional class improvement | baseline, 6 months follow-up, 12 months follow-up
  Secondary endpoint is bifocal stimulation therapy clinical response defined by New York Heart Association functional class scale, that is a method defining functional status of patients with heart failure. It has four categories (scale range: class 1-2-3-4) based on how much patients are limited during physical activity. Class 1 is the better outcome:no limitation of physical activity and ordinary physical activity does not cause fatigue, palpitation, dyspnea. Class 2: slight limitation of physical activity,comfortable at rest;ordinary physical activity results in fatigue, palpitation, dyspnea. Class 3:marked limitation of physical activity;comfortable at rest;less than ordinary activity causes fatigue, palpitation, or dyspnea. Class 4 is the worst outcome:unable to carry on any physical activity without discomfort; HF symptoms at rest and physical activity increases discomfort.
Left ventricular ejection fraction (LVEF) improvement major or equal than 25% compared to baseline and VVI mode, as evaluated by echocardiography. | baseline, 6 months follow-up, 12 months follow-up
  Secondary endpoint is bifocal stimulation therapy response defined by improvement of LVEF, as assessed by echocardiography. Specifically an improvement, obtained during bifocal stimulation in comparison to baseline and VVI-mode will be registered and would be significative for a cut off major or equal than 25%.
Left ventricular telesystolic volume reduction major or equal than 15% compared to baseline and VVI mode, as assessed by echocardiography. | baseline, 6 months follow-up, 12 months follow-up
  Secondary endpoint is bifocal stimulation therapy response defined by reduction major or equal than 15% of left ventricular telesystolic volume , as assessed by echocardiography

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital "Maggiore della Carità", Division of Cardiology, Novara, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nery PB, Ha AC, Keren A, Birnie DH. Cardiac resynchronization therapy in patients with left ventricular systolic dysfunction and right bundle branch block: a systematic review. Heart Rhythm. 2011 Jul;8(7):1083-7. doi: 10.1016/j.hrthm.2011.01.041. Epub 2011 Feb 4. PMID 21300176
- [Result] Barold SS, Audoglio R, Ravazzi PA, Diotallevi P. Is bifocal right ventricular pacing a viable form of cardiac resynchronization? Pacing Clin Electrophysiol. 2008 Jul;31(7):789-94. doi: 10.1111/j.1540-8159.2008.01093.x. No abstract available. PMID 18684274
- [Result] Res JC, Bokern MJ, de Cock CC, van Loenhout T, Bronzwaer PN, Spierenburg HA; BRIGHT Investigators. The BRIGHT study: bifocal right ventricular resynchronization therapy: a randomized study. Europace. 2007 Oct;9(10):857-61. doi: 10.1093/europace/eum147. Epub 2007 Aug 7. PMID 17684064